CLINICAL TRIAL: NCT07363382
Title: The Value of Gastrin-Releasing Peptide Receptor (GRPR) PET Imaging for Diagnosis and Staging in Prostate Cancer
Brief Title: The Value of GRPR PET Imaging for Diagnosis and Staging in Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-GRPR PET Imaging
Record Dates: First submitted 2026-01-16; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer (Adenocarcinoma)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 68Ga-G21 PET imaging (Experimental): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-G21. Tracer of 68Ga-G21 will be used to image lesions of prostate cancer by PET imaging.
  Interventions: Drug: 68Ga-G21
- 68Ga-G23 PET imaging (Experimental): Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-G23. Tracer of 68Ga-G23 will be used to image lesions of prostate cancer by PET imaging.
  Interventions: Drug: 68Ga-G23

INTERVENTIONS:
Drug: 68Ga-G21 — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-G21. Tracer of 68Ga-G21 will be used to image lesions of prostate cancer by PET imaging.
  Arms: 68Ga-G21 PET imaging
Drug: 68Ga-G23 — Intravenous injection of one dosage of 111-148 MBq (3-4 mCi) 68Ga-G23. Tracer of 68Ga-G23 will be used to image lesions of prostate cancer by PET imaging.
  Arms: 68Ga-G23 PET imaging

SUMMARY:
The gastrin-releasing peptide receptor (GRPR) is highly expressed in prostate cancer (77%-100%). Numerous studies have confirmed that GRPR PET imaging has emerged as a significant molecular imaging modality in prostate cancer, particularly serving as a complementary tool to PSMA PET for addressing cases with negative or insufficient PSMA expression. It demonstrates substantial value in initial staging (especially in intermediate- and high-risk patients), detecting sites of biochemical recurrence, assessing metastatic lesions (notably in mCRPC), and guiding treatment decisions. 68Ga-G21 and 68Ga-G23 are two novel molecular probes targeting GRPR. This study aims to evaluate their biodistribution and diagnostic performance in prostate cancer and compare them with 68Ga-PSMA-11 PET imaging.

DETAILED DESCRIPTION:
The gastrin-releasing peptide receptor (GRPR), also known as the bombesin receptor subtype BB2, is a G protein-coupled receptor containing seven transmembrane domains. Its endogenous ligand, gastrin-releasing peptide (GRP), exhibits high homology at the C-terminal peptide sequence with bombesin (BBN), a 14-amino-acid peptide derived from amphibians. GRP regulates a series of physiological processes including cell proliferation, differentiation, and metabolism by activating GRPR and its downstream phospholipase C signaling pathway. Studies have shown that GRPR is highly expressed in various malignant tumors and their metastases, such as gastrinoma (100%), prostate cancer (77%-100%), glioma (85%), gastrointestinal stromal tumors (84%), and breast cancer (62%-71.9%), and is closely associated with tumor growth, invasion, and metastasis. Owing to its widespread and high expression across multiple tumor types, GRPR has emerged as a pan-cancer target of significant clinical value, demonstrating strong potential for applications in the fields of precise tumor diagnosis and targeted therapy. Numerous studies have confirmed that GRPR PET imaging has emerged as a significant molecular imaging modality in prostate cancer, particularly serving as a complementary tool to PSMA PET for addressing cases with negative or insufficient PSMA expression. It demonstrates substantial value in initial staging (especially in intermediate- and high-risk patients), detecting sites of biochemical recurrence, assessing metastatic lesions (notably in mCRPC), and guiding treatment decisions. 68Ga-G21 and 68Ga-G23 are two novel molecular probes targeting GRPR. This study aims to evaluate their biodistribution and diagnostic performance in prostate cancer and compare them with 68Ga-PSMA-11 PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated prostate cancer patients;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Imaging Emergent Adverse Events | From enrollment till 7 days safety follow-up
  The distribution of adverse events (AE) will be done via the analysis of frequencies for imaging emergent Adverse Event, through the monitoring of relevant clinical and laboratory safety parameters.
Dosimetry data | through study completion, an average of 3 months
  Calculate the absorbed dose of 68Ga-G21 and 68Ga-G23 in normal organs.

SECONDARY OUTCOMES:
Diagnostic value | through study completion, an average of 3 months
  Sensitivity and Specificity of 68Ga-G21 and 68Ga-G23 PET imaging for prostate cancer in comparison with 68Ga-PSMA-11 PET imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China